CLINICAL TRIAL: NCT00960609
Title: Communicating Veins Between Adjacent Hepatic Veins: Rare, Exceptional or Frequent? An Intra-operative Ultrasound Study
Brief Title: Communicating Veins Between Adjacent Hepatic Veins: an Intra-operative Ultrasound Study
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Guido Torzilli, MD, PhD, University of Milan, Istituto Clinico Humanitas IRCCS
Other Study IDs: CV-HV
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Liver Tumors
Keywords: Communicating veins; hepatic venous anastomosis; intra-operative ultrasonography; hepatic resection; hepatic neoplasm; Primary and metastatic liver tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- caval confluence HV involvement: Patients carriers of primary or metastatic tumour with direct contact or invasion of one HV at the caval confluence.
  Interventions: Procedure: Ultrasound guided liver resection

INTERVENTIONS:
Procedure: Ultrasound guided liver resection

SUMMARY:
The search for communicating veins (CVs) between adjacent hepatic veins (HVs) has drawn its rationale from living donor liver transplantation (LDLT). Parenchymal sparing procedures although HVs are resected suggest that probably their presence is underestimated.

Taking profit from new improvements in ultrasound technology the investigators aim to better estimate the rate of CVs in a consecutive series of patients in whom resection of one HV at caval confluence is needed.

DETAILED DESCRIPTION:
The search for communicating veins (CVs) between adjacent hepatic veins (HVs) has drawn its rationale from the need of reducing the risk of incomplete blood outflow in the medial portion of the hemiliver without the middle hepatic vein (MHV) in living donor liver transplantation (LDLT). However, only 24% of patients seems having CVs based on the findings of color-Doppler intraoperative ultrasound (CD-IOUS) exploration. On the other hand the safety of parenchymal sparing procedure despite HV resection let suppose that CVs are probably more frequent than expected.

Certainly, better in vivo knowledge of the rate of CVs and their direct detection would consolidate and probably further expand parenchymal sparing techniques. Taking profit from new advancements in ultrasound technology we have carried out the present study with the aim of better estimating the rate of CVs in a consecutive series of patients in whom resection of one HV at caval confluence was needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for being enrolled in the present study were those carriers of primary or metastatic tumour with direct contact or invasion of one HV at the caval confluence.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary and metastatic liver tumors addressed to surgical treatment
Sampling Method: Probability Sample
Dates: Start 2008-01

PRIMARY OUTCOMES:
First outcome was the rate of CVs detectable with e-flow IOUS along clamping of the HV for which resection could be needed.

SECONDARY OUTCOMES:
Secondary outcome was safety (morbidity, mortality, blood loss, blood transfusions) of the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, IRCCS, Rozzano, Milano, Italy

REFERENCES:
- [Background] Torzilli G, Procopio F, Botea F, Marconi M, Del Fabbro D, Donadon M, Palmisano A, Spinelli A, Montorsi M. One-stage ultrasonographically guided hepatectomy for multiple bilobar colorectal metastases: a feasible and effective alternative to the 2-stage approach. Surgery. 2009 Jul;146(1):60-71. doi: 10.1016/j.surg.2009.02.017. PMID 19541011
- [Background] Torzilli G, Donadon M, Marconi M, Palmisano A, Del Fabbro D, Spinelli A, Botea F, Montorsi M. Hepatectomy for stage B and stage C hepatocellular carcinoma in the Barcelona Clinic Liver Cancer classification: results of a prospective analysis. Arch Surg. 2008 Nov;143(11):1082-90. doi: 10.1001/archsurg.143.11.1082. PMID 19015467
- [Background] Torzilli G, Donadon M, Marconi M, Botea F, Palmisano A, Del Fabbro D, Procopio F, Montorsi M. Systematic extended right posterior sectionectomy: a safe and effective alternative to right hepatectomy. Ann Surg. 2008 Apr;247(4):603-11. doi: 10.1097/SLA.0b013e31816387d7. PMID 18362622
- [Background] Torzilli G, Donadon M, Palmisano A, Del Fabbro D, Spinelli A, Makuuchi M, Montorsi M. Back-flow bleeding control during resection of right-sided liver tumors by means of ultrasound-guided finger compression of the right hepatic vein at its caval confluence. Hepatogastroenterology. 2007 Jul-Aug;54(77):1364-7. PMID 17708255
- [Background] Torzilli G, Montorsi M, Del Fabbro D, Palmisano A, Donadon M, Makuuchi M. Ultrasonographically guided surgical approach to liver tumours involving the hepatic veins close to the caval confluence. Br J Surg. 2006 Oct;93(10):1238-46. doi: 10.1002/bjs.5321. PMID 16953487
- [Background] Sano K, Makuuchi M, Miki K, Maema A, Sugawara Y, Imamura H, Matsunami H, Takayama T. Evaluation of hepatic venous congestion: proposed indication criteria for hepatic vein reconstruction. Ann Surg. 2002 Aug;236(2):241-7. doi: 10.1097/00000658-200208000-00013. PMID 12170030